CLINICAL TRIAL: NCT02851680
Title: Prospective Study on the Interest of ß 1-3 D Glucan Assays in Screening for the Onset of Invasive Aspergillosis in Neutropenic Patients With Acute Leukaemia.
Brief Title: Interest of ß 1-3 D Glucan Assays in Screening for the Onset of Invasive Aspergillosis in Neutropenic Patients With Acute Leukaemia.
Acronym: BETA GLUCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: DALLE 2013
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-06

CONDITIONS: Invasive Fungal Infections
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Blood Specimen Collection

ARMS (2):
- Fongitell test (Experimental)
  Interventions: Biological: blood samples
- serum galactomannan (Active Comparator)
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples

SUMMARY:
In the context of screening for infectious fungal diseases in patients with malignant haemopathy, and particularly patients with acute leukaemia, the investigator aims to evaluate the performance of an already commercialized but little used serum screening test (Fungitell® test) and to determine its place in the management strategy for invasive aspergillosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been informed about the study
* Patients over 18 years
* patients with acute myeloblastic leukaemia (AML) or lymphoblastic leukaemia (ALL) who have undergone cytotoxic chemotherapy with curative intent

Exclusion Criteria:

* Adults under guardianship
* Patients without national health insurance cover
* Pregnant or breast-feeding women
* allografts and autografts of Haematopoietic Stem Cells (HSC)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Comparison of the results of the 1-3 ß D glucan serum assay obtained with the Fungitell® test and the test currently used (in terms of specificity, sensitivity, negative predictive value and positive predictive value | 8 to 10 assays over 4 to 5 weeks of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France